CLINICAL TRIAL: NCT02476617
Title: An Exploratory Study to Evaluate Immune Restoration Following Removal of Viral Antigen in Treatment-Naïve and Treatment-Experienced Adults With Genotype (GT) 1a Chronic Hepatitis C Virus (HCV) Infection Administered Ombitasvir/ ABT-450/Ritonavir With Dasabuvir and Ribavirin (RBV) for 12 Weeks
Brief Title: Ombitasvir/ABT-450 (Paritaprevir)/Ritonavir With Dasabuvir and Ribavirin (RBV) in Treatment Naive and Treatment Experienced Genotype 1a Hepatitis C Virus Infected Adults
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M14-243
Record Dates: First submitted 2015-06-17; First posted 2015-06-19 (Estimated); Results first posted 2017-09-05 (Actual); Last update posted 2017-10-03 (Actual); Status verified 2017-08

CONDITIONS: Chronic Hepatitis C; Hepatitis C (HCV); Hepatitis C Genotype 1a
Keywords: Treatment naive; Interferon free; HCV; Chronic Hepatitis C; Hepatitis C Genotype 1a; Hepatitis C; pegylated-interferon (pegIFN)/ribavirin (RBV) experienced
MeSH Terms: conditions — Hepatitis C, Chronic; Hepatitis C | interventions — ombitasvir; dasabuvir; Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Ombitasvir/paritaprevir/ritonavir + dasabuvir + RBV (Experimental): Ombitasvir/paritaprevir/ritonavir (25 mg/150 mg/100 mg once daily [QD]) + dasabuvir (250 mg twice daily [BID]) + weight based Ribavirin (RBV; dosed 1,000 or 1,200 mg daily divided BID)
  Interventions: Drug: ombitasvir/paritaprevir/ritonavir; Drug: dasabuvir; Drug: ribavirin

INTERVENTIONS:
Drug: ombitasvir/paritaprevir/ritonavir — ombitasvir/ABT-450/ritonavir tablets
  Other Names: ABT-267/ABT-450/ritonavir
Drug: dasabuvir — dasabuvir tablets
  Other Names: ABT-333
Drug: ribavirin — ribavirin tablets

SUMMARY:
A study to evaluate immune restoration following removal of viral antigen in non-cirrhotic hepatitis C virus (HCV) genotype (GT) 1a treatment-naïve and pegylated-interferon (pegIFN)/ribavirin (RBV) treatment-experienced adults receiving treatment with ombitasvir/paritaprevir/ritonavir and dasabuvir coadministered with ribavirin (RBV) for 12 weeks.

DETAILED DESCRIPTION:
A study to evaluate the role of ombitasvir/paritaprevir/ritonavir and dasabuvir coadministered with RBV treatment leading to sustained virologic response 12 weeks post-dosing (SVR12) on the changes from baseline in IFN-stimulated gene (ISG) expression in peripheral blood mononucleated cells (PBMCs) in HCV GT 1a-infected adult participants.

ELIGIBILITY:
Inclusion Criteria:

1. Screening laboratory result indicating hepatitis C viral (HCV) genotype (GT) 1a infection.
2. Chronic HCV infection.
3. Participants must be non-cirrhotic.
4. Participants must be treatment-naïve or have documentation that they were adherent to prior pegIFN/RBV combination therapy and meet the criteria of prior pegylated-interferon (pegIFN)/ribavirin (RBV) treatment failure.
5. Participants must meet specific human leukocyte antigen (HLA) allele requirements.

Exclusion Criteria:

1. Women who are pregnant or breastfeeding.
2. Positive test result for hepatitis B surface antigen (HBsAg) or anti-human immunodeficiency virus antibody (HIV Ab) positive immunoassay.
3. Clinically significant abnormalities or co-morbidities, other than HCV infection, that make the subject unsuitable for this study or treatment.
4. Current enrollment in another interventional clinical study, previous enrollment in this study, prior or current use of any investigational or commercially available anti-HCV agents other than pegIFN or RBV (including previous exposure to paritaprevir, ombitasvir, or dasabuvir), or receipt of any investigational product within 6 weeks prior to study drug administration.
5. History of solid organ transplant.
6. Screening laboratory analysis that shows abnormal results.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2015-06; Primary Completion 2016-08 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Emily Dumas, PhD, Study Director — AbbVie

REFERENCES:
- [Derived] Cui A, Li B, Wallace MS, Gonye ALK, Oetheimer C, Patel H, Tonnerre P, Holmes JA, Lieb D, Yao BS, Ma A, Roberts K, Damasio M, Chen JH, Piou D, Carlton-Smith C, Brown J, Mylvaganam R, Hon Fung JM, Sade-Feldman M, Aneja J, Gustafson J, Epstein ET, Salloum S, Brisac C, Thabet A, Kim AY, Lauer GM, Hacohen N, Chung RT, Alatrakchi N. Single-cell atlas of the liver myeloid compartment before and after cure of chronic viral hepatitis. J Hepatol. 2024 Feb;80(2):251-267. doi: 10.1016/j.jhep.2023.02.040. Epub 2023 Mar 25. PMID 36972796
- [Derived] Tonnerre P, Wolski D, Subudhi S, Aljabban J, Hoogeveen RC, Damasio M, Drescher HK, Bartsch LM, Tully DC, Sen DR, Bean DJ, Brown J, Torres-Cornejo A, Robidoux M, Kvistad D, Alatrakchi N, Cui A, Lieb D, Cheney JA, Gustafson J, Lewis-Ximenez LL, Massenet-Regad L, Eisenhaure T, Aneja J, Haining WN, Chung RT, Hacohen N, Allen TM, Kim AY, Lauer GM. Differentiation of exhausted CD8+ T cells after termination of chronic antigen stimulation stops short of achieving functional T cell memory. Nat Immunol. 2021 Aug;22(8):1030-1041. doi: 10.1038/s41590-021-00982-6. Epub 2021 Jul 26. PMID 34312544

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The intent-to-treat (ITT) population consisted of all enrolled participants who received at least one dose of study drug.
Period: Overall Study
Arm/Group | Ombitasvir/Paritaprevir/Ritonavir + Dasabuvir + RBV
Started | 25
Completed | 23
Not Completed | 2
Not completed — Adverse Event | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Population: Safety and demographic analyses were performed on safety population, which is the same as the ITT population.
Groups:
- Ombitasvir/Paritaprevir/Ritonavir + Dasabuvir + RBV: Ombitasvir/paritaprevir/ritonavir (25 mg/150 mg/100 mg QD) + dasabuvir (250 mg BID) + weight based Ribavirin (RBV; dosed 1,000 or 1,200 mg daily divided BID)
Arm/Group | Ombitasvir/Paritaprevir/Ritonavir + Dasabuvir + RBV
Number analyzed (Participants) | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.8 (12.61)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 19

OUTCOME MEASURES:

1. Primary Outcome: Change in Interferon (IFN)-Stimulated Genes (ISG) Expression in Peripheral Blood Mononucleated Cells (PBMCs) for Participants Achieving SVR12
Description: The changes from week 0 to post-treatment (PT) week 12 in key ISG expression in PBMCs for participants achieving sustained virologic response 12 weeks PT (SVR12) where SVR12 was defined as hepatitis C virus ribonucleic acid (HCV RNA) level less than the lower limit of quantification (<LLOQ) 12 weeks after the last dose of study drug. For each key ISG, fold change was defined as the ratio of the difference between PT Week 12 and baseline expressions over the baseline expression.
Time Frame: Week 0 to Post-Treatment Week 12
Population: All participants who achieved SVR12 and had both baseline and post-baseline value at Post-Treatment Week 12 were included in this analyses..
Measure: Mean (Standard Deviation); unit: Fold change
Arm/Group | Ombitasvir/Paritaprevir/Ritonavir + Dasabuvir + RBV
Number analyzed (Participants) | 21
Fold change
  CXCL10 | -0.464 (0.6143)
  ISG15 | -0.148 (0.7458)
  CXCL11 | -0.611 (0.3090)
  MX1 | -0.399 (0.3013)
  IFI27 | -0.462 (0.4624)
  OAS2 | -0.168 (0.5168)
  DDX60 | -0.016 (0.5696)
  IFIT3 | -0.543 (0.3350)
  IFI44 | -0.467 (0.2569)
  STAT1 | -0.301 (0.3430)
  CXCL9 | -0.552 (0.2816)
  IFIT1 | -0.440 (0.4441)
  HERC5 | -0.358 (0.2827)
  IRF7 | -0.171 (0.4273)
  OAS1 | 0.284 (1.4668)
  PLSCR1: number analyzed (Participants) | 20
  PLSCR1 | -0.255 (0.3688)
  IRF9 | -0.205 (0.2809)
  IFIH1 | -0.321 (0.3213)
  TRIM14 | 0.022 (0.5282)
  IRF1 | -0.130 (0.6497)
  IRF3 | 0.044 (0.6307)
  STAT2 | -0.051 (0.5762)
  IFNG | 0.516 (1.4653)
  IFNL1 | -0.361 (0.3753)
  IFNL2 | -0.199 (0.7031)
  IFNL3 | -0.205 (0.4306)
  IFNL4 | -0.228 (0.7298)
  IFNGR1 | -0.046 (0.3008)
  ADAR | -0.212 (0.2314)
  ALG10 | -0.083 (0.7491)
  BCHE | -0.101 (0.5739)
  CCL2 | 0.200 (1.5071)
  CCL4 | 0.638 (1.7396)
  CD163 | 0.556 (2.7478)
  CXCL5: number analyzed (Participants) | 19
  CXCL5 | 1.085 (2.7539)
  CXCR3 | 0.308 (0.5236)
  DDIT4 | 0.029 (1.2134)
  DDX58 | 0.388 (1.2231)
  DPP4 | 0.869 (1.5730)
  EIF2AK2 | -0.317 (0.2521)
  GBP1 | -0.288 (0.4421)
  GCKR | 0.009 (0.5267)
  GUCY1B3 | 0.350 (0.7909)
  HELZ2 | -0.232 (0.5124)
  HERC6 | -0.074 (0.3294)
  IFI35 | -0.023 (0.6428)
  IFI44L: number analyzed (Participants) | 20
  IFI44L | -0.554 (0.4068)
  IFI6 | -0.464 (0.3010)
  IFIT2 | -0.365 (0.4118)
  IFIT5 | -0.291 (0.2085)
  IFITM1 | -0.066 (0.3696)
  IFITM2 | 0.158 (0.7905)
  IFITM3 | -0.423 (0.3313)
  IFNA | -0.202 (0.5037)
  IFNB | -0.167 (0.4427)
  IL10 | 0.202 (0.8216)
  IL18 | -0.078 (0.2695)
  IRF2: number analyzed (Participants) | 20
  IRF2 | 0.311 (1.0487)
  ISG20 | 0.156 (1.0071)
  MAP3K14 | -0.072 (0.2983)
  MOV10 | -0.185 (0.4048)
  MS4A4A: number analyzed (Participants) | 20
  MS4A4A | -0.005 (0.7458)
  MX2 | -0.101 (0.6188)
  MYST1 | -0.057 (0.2404)
  NOS2A: number analyzed (Participants) | 20
  NOS2A | 0.249 (0.8288)
  NT5C3 | 0.017 (0.3577)
  OASL | -0.233 (0.6984)
  PPP3CB | 0.011 (0.1956)
  RNASEL | 0.395 (0.9973)
  RSAD2 | -0.406 (0.3202)
  SLC27A2: number analyzed (Participants) | 20
  SLC27A2 | 0.022 (0.9149)
  SOCS1 | 1.313 (3.5778)
  SOCS3 | 0.025 (1.1773)
  USP18 | -0.288 (0.3092)

ADVERSE EVENTS:
Time Frame: Treatment-emergent AEs (TEAEs) and treatment-emergent SAEs (TESAEs) were collected from first dose of study drug until 30 days after the last dose of study drug (up to 16 weeks).
Description: TEAEs and TESAEs are defined as any adverse event (AE) with an onset date that is after the first dose of study drug until 30 days after the last dose of study drug and were collected whether elicited or spontaneously reported by the participant.
Groups:
- Ombitasvir/Paritaprevir/Ritonavir + Dasabuvir + RBV: Arm/Group Description: Ombitasvir/paritaprevir/ritonavir (25 mg/150 mg/100 mg QD) + dasabuvir (250 mg BID) + weight based Ribavirin (RBV; dosed 1,000 or 1,200 mg daily divided BID)
Arm/Group | Ombitasvir/Paritaprevir/Ritonavir + Dasabuvir + RBV
Serious Adverse Events (participants affected / at risk) | 2/25
Other Adverse Events (participants affected / at risk) | 24/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ombitasvir/Paritaprevir/Ritonavir + Dasabuvir + RBV (N=25)
OVERDOSE (Injury, poisoning and procedural complications) | 1
ANXIETY (Psychiatric disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ombitasvir/Paritaprevir/Ritonavir + Dasabuvir + RBV (N=25)
EXCESSIVE CERUMEN PRODUCTION (Ear and labyrinth disorders) | 1
VERTIGO (Ear and labyrinth disorders) | 1
ABDOMINAL DISCOMFORT (Gastrointestinal disorders) | 3
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 1
CONSTIPATION (Gastrointestinal disorders) | 4
DIARRHOEA (Gastrointestinal disorders) | 5
DYSPEPSIA (Gastrointestinal disorders) | 4
DYSPHAGIA (Gastrointestinal disorders) | 1
ERUCTATION (Gastrointestinal disorders) | 1
FAECES DISCOLOURED (Gastrointestinal disorders) | 2
HAEMATOCHEZIA (Gastrointestinal disorders) | 1
IRRITABLE BOWEL SYNDROME (Gastrointestinal disorders) | 1
NAUSEA (Gastrointestinal disorders) | 9
RETCHING (Gastrointestinal disorders) | 2
VOMITING (Gastrointestinal disorders) | 3
ASTHENIA (General disorders) | 3
CHEST DISCOMFORT (General disorders) | 1
CHEST PAIN (General disorders) | 1
CYST (General disorders) | 1
FATIGUE (General disorders) | 16
FEELING JITTERY (General disorders) | 1
MALAISE (General disorders) | 3
PAIN (General disorders) | 1
PERIPHERAL SWELLING (General disorders) | 2
BILIARY DILATATION (Hepatobiliary disorders) | 1
HYPERSENSITIVITY (Immune system disorders) | 2
BRONCHITIS (Infections and infestations) | 1
EAR INFECTION (Infections and infestations) | 1
GASTROENTERITIS VIRAL (Infections and infestations) | 2
HERPES ZOSTER (Infections and infestations) | 1
INFECTED DERMAL CYST (Infections and infestations) | 1
INFLUENZA (Infections and infestations) | 2
NASOPHARYNGITIS (Infections and infestations) | 3
SINUSITIS (Infections and infestations) | 1
TOOTH INFECTION (Infections and infestations) | 1
HAND FRACTURE (Injury, poisoning and procedural complications) | 1
JOINT DISLOCATION (Injury, poisoning and procedural complications) | 1
LIGAMENT SPRAIN (Injury, poisoning and procedural complications) | 1
MUSCLE STRAIN (Injury, poisoning and procedural complications) | 1
ROAD TRAFFIC ACCIDENT (Injury, poisoning and procedural complications) | 1
BLOOD BILIRUBIN INCREASED (Investigations) | 4
CREATININE RENAL CLEARANCE DECREASED (Investigations) | 1
HAEMATOCRIT DECREASED (Investigations) | 1
HAEMOGLOBIN DECREASED (Investigations) | 4
DECREASED APPETITE (Metabolism and nutrition disorders) | 3
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 2
ARTHRITIS (Musculoskeletal and connective tissue disorders) | 1
BACK PAIN (Musculoskeletal and connective tissue disorders) | 1
FLANK PAIN (Musculoskeletal and connective tissue disorders) | 1
MUSCULOSKELETAL STIFFNESS (Musculoskeletal and connective tissue disorders) | 1
MYALGIA (Musculoskeletal and connective tissue disorders) | 3
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 1
SPINAL COLUMN STENOSIS (Musculoskeletal and connective tissue disorders) | 1
BURNING SENSATION (Nervous system disorders) | 1
DIZZINESS (Nervous system disorders) | 4
DYSGEUSIA (Nervous system disorders) | 1
HEADACHE (Nervous system disorders) | 6
HYPOAESTHESIA (Nervous system disorders) | 2
LOSS OF CONSCIOUSNESS (Nervous system disorders) | 1
PARAESTHESIA (Nervous system disorders) | 1
POOR QUALITY SLEEP (Nervous system disorders) | 2
RESTLESS LEGS SYNDROME (Nervous system disorders) | 2
SYNCOPE (Nervous system disorders) | 1
ANXIETY (Psychiatric disorders) | 4
DEPRESSION (Psychiatric disorders) | 1
INSOMNIA (Psychiatric disorders) | 6
IRRITABILITY (Psychiatric disorders) | 4
MOOD SWINGS (Psychiatric disorders) | 1
TACHYPHRENIA (Psychiatric disorders) | 1
CHROMATURIA (Renal and urinary disorders) | 1
NEPHROLITHIASIS (Renal and urinary disorders) | 1
COUGH (Respiratory, thoracic and mediastinal disorders) | 1
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 4
HAEMOPTYSIS (Respiratory, thoracic and mediastinal disorders) | 1
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 2
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 1
HYPERHIDROSIS (Skin and subcutaneous tissue disorders) | 1
PRURITUS (Skin and subcutaneous tissue disorders) | 3
PSORIASIS (Skin and subcutaneous tissue disorders) | 1
RASH (Skin and subcutaneous tissue disorders) | 3
SKIN IRRITATION (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.